CLINICAL TRIAL: NCT06764030
Title: A Pilot Feasibility Study of a Patient-Directed Computerized Intervention to Address Reproductive Coercion
Brief Title: A Patient-Directed Computerized Intervention to Address Reproductive Coercion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Yasamin Yoko Kusunoki, Associate Professor, University of Michigan
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HUM00259457; R21HD107619 (NIH)
Record Dates: First submitted 2024-12-01; First posted 2025-01-08 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Feasibility Pilot Study

STUDY DESIGN:
Intervention Model Description: The intervention group will interact with BRIDGES in addition to receiving standard of care while the control group will receive standard of care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BRIDGES plus standard of care (Experimental)
  Interventions: Other: Educational web-based application
- Standard of care (No Intervention)

INTERVENTIONS:
Other: Educational web-based application — BRIDGES is a patient-directed computerized universal education on RC that is delivered within the FP setting, and that does not require the patient to disclose RC experiences to learn about RC.
  Arms: BRIDGES plus standard of care

SUMMARY:
The goal of this clinical trial is to evaluate the feasibility and acceptability of "BRIDGES" (Building Reproductive Decision-Making, Empowerment, & Support), a new patient-directed educational website (bridges4support.org). BRIDGES aims to improve family planning (FP) patients' understanding of reproductive coercion (RC) and harm-reduction strategies, as well as their ability to discuss RC-related issues with healthcare providers if they so choose. Designed to be integrated into routine FP clinical care and pre-visit materials, this brief (5-10 minute) educational website includes 1) education on reproductive coercion and (un)healthy relationships, 2) harm-reduction and safety planning strategies, and 3) patient activation messages to encourage patients to actively engage with their healthcare provider. Four study clinics were selected from Planned Parenthood of Michigan (PPMI) clinics based on patient volume and number of clinics. Two of the four chosen clinics will be randomly assigned to receive BRIDGES, with 40 participants per clinic, and the other two clinics will be randomly assigned to receive the standard of care, also with 40 participants per clinic. Control clinics will receive the standard of care, which includes the typical support and counseling provided at these centers for FP patients, and the intervention clinics will receive BRIDGES plus standard of care. Research staff will recruit FP patients ages 18-29 (N=160) through patient portal messages. Participants will complete online, self-directed Qualtrics surveys at three time points: pre-appointment, post-appointment, and 3-months. Survey data will be used to assess differences in patient knowledge, self-efficacy, and behavior between patients attending intervention clinics and patients attending control FP clinics (i.e., receiving standard-of-care FP services). Feasibility, implementation, and pilot outcome data will be used to further refine the intervention towards the goal of conducting a future larger-scale study of BRIDGES within FP clinics.

ELIGIBILITY:
Inclusion Criteria:

* Family planning patients at study clinics, including women, transgender men, non-binary, and other gender-diverse people
* Ages 18-29
* Able to participate in English
* Has an upcoming birth control appointment (telemedicine or in-clinic) scheduled at a study clinic during the enrollment period (November 2024-June 2025). Appointments must be scheduled for at least 24 hours after study enrollment.
* Has access to PPMI MyChart (i.e., study clinic patient portal)
* Participants who complete the Pre-Appointment Survey and attend the scheduled birth control appointment or a rescheduled (up to 3x) appointment are eligible for the Post-Appointment Survey
* Participants who complete the Pre-Appointment Survey are eligible for the 3-Month Survey, regardless of whether they complete the Post-Appointment Survey

Exclusion Criteria:

* Previously exposed to the intervention (e.g., participated in user testing during September and October 2024)
* Does not have a valid email address

Ages: 18 Years to 29 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 156 (Actual)
Dates: Start 2024-11-18 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Level of agreement that the BRIDGES website was acceptable | Up to five days after appointment
  In a self-administered survey, patients at the treatment clinic are asked the extent to which they agree with the following statements: The BRIDGES website is an acceptable way to learn about each of the following (reproductive coercion, birth control methods that other people are less able to control, things to discuss with a healthcare provider, resources, and use of the patient portal for the invitation to the study). Reponse options for each statement ranged from strongly disagree (1) to strongly agree (5) such that a higher score would signify agreement with the statement.
Level of agreement that the user liked BRIDGES | Up to five days after appointment
  In a self-administered survey, patients at the treatment clinic are asked the extent to which they agree with the following statement: I like the bridges website. Response options for each statement ranged from strongly disagree (1) to strongly agree (5) such that a higher score would signify agreement with the statement.
Level of agreement that BRIDGES was helpful | Up to five days after appointment
  In a self-administered survey, patients at the treatment clinic are asked the extent to which they agree with the following statement: Overall, the BRIDGES website helped me. Response options for each statement ranged from strongly disagree (1) to strongly agree (5) such that a higher score would signify agreement with the statement.
Level of agreement that the user was comfortable using BRIDGES | Up to five days after appointment
  In a self-administered survey, patients at the treatment clinic are asked the extent to which they agree with the following statement: I felt uncomfortable when viewing the BRIDGES website. Response options for each statement ranged from strongly disagree (1) to strongly agree (5) such that a higher score would signify agreement with the statement.
Level of agreement that the user felt safe using BRIDGES | Up to five days after appointment
  In a self-administered survey, patients at the treatment clinic are asked the extent to which they agree with the following statement: I felt unsafe when viewing the BRIDGES website. Response options for each statement ranged from strongly disagree (1) to strongly agree (5) such that a higher score would signify agreement with the statement.
Level of agreement that BRIDGES was easy to use | Up to five days after appointment
  In a self-administered survey, patients at the treatment clinic are asked the extent to which they agree with the following statement: The BRIDGES website was easy to use. Response options for each statement ranged from strongly disagree (1) to strongly agree (5) such that a higher score would signify agreement with the statement.
Level of agreement that the BRIDGES website helped them talk to their healthcare provider about their intimate relationships | Up to five days after appointment
  In a self-administered survey, patients at the treatment clinic are asked the extent to which they agree with the following statement: The BRIDGES website helped me talk to my healthcare provider about my intimate relationships. Response options for each statement ranged from strongly disagree (1) to strongly agree (5) such that a higher score would signify agreement with the statement.
Level of agreement that the BRIDGES website helped them talk to their healthcare provider about their preferred birth control method | Up to five days after appointment
  In a self-administered survey, patients at the treatment clinic are asked the extent to which they agree with the following statement: The BRIDGES website helped me talk to my healthcare provider about my preferred birth control method. Response options for each statement ranged from strongly disagree (1) to strongly agree (5) such that a higher score would signify agreement with the statement.
Level of agreement that the BRIDGES website helped them choose a birth control method that works best for them | Up to five days after appointment
  In a self-administered survey, patients at the treatment clinic are asked the extent to which they agree with the following statement: The BRIDGES website helped me choose a birth control method that works best for me. Response options for each statement ranged from strongly disagree (1) to strongly agree (5) such that a higher score would signify agreement with the statement.
Level of agreement that the BRIDGES website influenced their decision about which birth control method they wanted | Up to five days after appointment
  In a self-administered survey, patients at the treatment clinic are asked the extent to which they agree with the following statement: The BRIDGES website influenced my decision about which birth control method I wanted. Response options for each statement ranged from strongly disagree (1) to strongly agree (5) such that a higher score would signify agreement with the statement.
Level of agreement that the BRIDGES website will help them talk to their friends and family about reproductive coercion | Up to five days after appointment
  In a self-administered survey, patients at the treatment clinic are asked the extent to which they agree with the following statement: The BRIDGES website will help me talk to my friends and family about reproductive coercion. Response options for each statement ranged from strongly disagree (1) to strongly agree (5) such that a higher score would signify agreement with the statement.
Level of agreement that the user would share the BRIDGES website with a friend or family member who needed support | Up to five days after appointment
  In a self-administered survey, patients at the treatment clinic are asked the extent to which they agree with the following statement: I would share the BRIDGES website with a friend or family member who needed support. Response options for each statement ranged from strongly disagree (1) to strongly agree (5) such that a higher score would signify agreement with the statement.
Level of agreement that the user would use the BRIDGES website if the user were not in the study | Up to five days after appointment
  In a self-administered survey, patients at the treatment clinic are asked the extent to which they agree with the following statement: If I was not in this research study, I would use the BRIDGES website. Response options for each statement ranged from strongly disagree (1) to strongly agree (5) such that a higher score would signify agreement with the statement.

SECONDARY OUTCOMES:
Knowledge about which birth control methods can be kept private | Pre-appointment
  In a self-administered survey, all patients are asked: Imagine you wanted to keep your birth control private. Which of the following birth control methods are more difficult for other people (like a partner) to mess with or control? (select all that apply). Seven types of birth control methods are provided. The correct answers include birth control implant, injectable birth control, intrauterine device, and sterilization. Incorrect answers include birth control pills, condoms, and withdrawal.
Change in knowledge about which birth control methods can be kept private | Three months after appointment
  In a self-administered survey, all patients are asked: Imagine you wanted to keep your birth control private. Which of the following birth control methods are more difficult for other people (like a partner) to mess with or control? (select all that apply). Seven types of birth control methods are provided. The correct answers include birth control implant, injectable birth control, intrauterine device, and sterilization. Incorrect answers include birth control pills, condoms, and withdrawal. A measure of change will be created by subtracting the number of correct methods 3 months after interacting with BRIDGES minus the number of correct methods before interacting with BRIDGES. A value of 0 will signify that knowledge remained the same; a positive value will signify that knowledge increased; a negative value will signify that knowledge decreased.
Knowledge about what reproductive coercion is | Pre-appointment
  In a self-administered survey, all patients are asked: TRUE or FALSE: Pressuring a partner to become pregnant when they don't want to be can be a sign of an unhealthy relationship. The correct answer is true.
Change in knowledge about what reproductive coercion is | Three months after appointment
  In a self-administered survey, all patients are asked: TRUE or FALSE: Pressuring a partner to become pregnant when they don't want to be can be a sign of an unhealthy relationship. The correct answer is true. A measure of change will be created that compares the answer to this question before and three months after interacting with BRIDGES. If the response is true at both time points or was false before and true after, it would signify an improvement in knowledge.
Knowledge about the role of healthcare providers | Pre-appointment
  In a self-administered survey, all patients are asked: TRUE or FALSE: Healthcare providers can support people who feel controlled in their reproductive decisions. The correct answer is true.
Change in knowledge about the role of healthcare providers | Three months after appointment
  In a self-administered survey, all patients are asked: TRUE or FALSE: Healthcare providers can support people who feel controlled in their reproductive decisions. The correct answer is true. A measure of change will be created that compares the answer to this question before and three months after their appointment. If the response is false before and true after, it would signify an improvement in knowledge.
Confidence in their ability to ask with their healthcare providers about issues related to reproductive coercion | Three months after appointment
  In a self-administered survey, all patients are asked the extent to which they agree with being confident in asking their healthcare provider about issues related to reproductive coercion. Response options for each statement ranged from strongly disagree (1) to strongly agree (5) such that a higher score would signify agreement with the statement. The responses to this question will be compared between the treatment and control.
Change in level of reproductive autonomy | Three months after appointment
  In a self-administered survey, all patients are asked about their level of reproductive autonomy based on a validated 14-item measure which included three subscales that encompass reproductive autonomy including communication, freedom from coercion, and decision-making. Mean scores were calculated for each subscale by adding the value of the response choice for each item on the subscale and dividing this value by the number of items on the subscale. Higher scores on each subscale represented higher levels of RA (score ranges from 0 to 14). A measure of change will be created that compares the answer to this question before and three months after their appointment.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No